CLINICAL TRIAL: NCT03042806
Title: Validation of a Questionnaire Evaluating the Physical Activities in COPD Patients: the Maugeri Physical Activity Questionnaire - MaPAct
Brief Title: Validation of a Questionnaire for Physical Activity in COPD: Maugeri Physical Activity Questionnaire (MaPAct)
Acronym: MaPAct
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elisabetta Zampogna (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Sponsor-Investigator, Elisabetta Zampogna, Principal Investigator, Fondazione Salvatore Maugeri
Organization: Fondazione Salvatore Maugeri (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ICSMaugeri
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: COPD
Keywords: Physical Activity; Questionnaire
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Other): COPD patients will be asked to fill in the Maugeri Physical Activity Questionnaire (MaPAct) to assess self perceived physical activity.
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — all the COPD patients will be ask to complete the questionnaire

SUMMARY:
Patients affected from Chronic Obstructive Pulmonary Disease (COPD) benefit from pulmonary rehabilitation in terms of exercise capacity, symptoms and health-related quality of life whereas the effect on physical activity is still not clear. Some studies have investigated the effect of exercise training on daily physical activity. However, there is considerable variability in study findings, data are discordant and the effect of exercise training on physical activity is unclear. There are probably a number of reasons to account for this.

First of all, the choice of the method for evaluating physical activity. Although direct observation, double-labelled water and calorimetry are considered the gold standard for assessing physical activity, they are too time consuming and expensive to be used in large population studies .The Physical Activity (PA) of patients with COPD can be assessed using questionnaires. A variety of questionnaires exist that capture different aspects of physical activity such as amount, type, intensity, symptom experience and limitations in the performance of ''activities of daily life''. Up to now, it still does not exist an instrument that evaluates the physical activity of COPD patients in Italian language that takes in account Italian people' lifestyle. Since this is strongly influenced by the environment, cultural and social conditions in which we live, it is essential to have an instrument specifically tailored for the population under study.

Aim of this study is to validate the Maugeri Physical Activity questionnaire (MaPAct) in COPD patients pointing to assess self-perceived physical activity.

DETAILED DESCRIPTION:
Methods The study will be approved by the Internal Review Board and Ethics Committee of the Salvatore Maugeri Foundation, Institute of Care and Scientific Research Rehabilitation of Tradate and Lumezzane, Italy and Malcantonese Hospital, Castelrotto, Switzerland. The procedures will be performed between September 2016 to September 2018.

Study design A team of experts, (1 pulmonologist, 1 bioengineer, 4 physiotherapists, 1 psychologist and 1 psychometrist) elaborated the instruments and defined the instructions to administer the MaPAct to self-evaluate the physical activity during daily life. This phase distinguishes three steps.

Subjects A total of 195 in-hospital patients (15 in a first step, 50 in a second step and 130 in the third) with diagnosis of COPD, will be enrolled. Will be excluded from the study all the patients that were hospitalized in the 30 days before admission, patients with degenerative neuromuscular disease, subjects with motor disabilities limiting ambulation, subjects with memory or comprehension problems, with dementia, Parkinson disease, and subjects that do not give their consent to the participation to the study. All subjects receive a consent informed.

Step 1 A focus group of 15 patients will be arranged and patients will be asked to fill in the preliminary version of the questionnaire and to offer their impression. In this pilot step patients will be also asked to discuss on the relevance for the study population and comprehensiveness of the items describing them generically as 'clear' or 'unclear', "appropriate" or "not appropriate" to themselves (16-17), the aim being to achieve consensus for each item. Where items were described as "not appropriate" or "unclear", participants should explain their reasons. Some items should be removed at this stage, or reworded if necessary. The objective was to include all items judged to be relevant to COPD patients. These items will form the Item Set.

Step 2 The patient-perceived comprehensibility will be tested on a sample of 50 patients. Patients will be asked to rank their perceived comprehensibility of the questionnaire on a 4-point Likert scale, between 0 and 3 (0 =Easy, 1 =Quite easy, 2 = Quite difficult, and 3 = Difficult). Some items should be removed at this stage, or reworded if necessary.

Step 3 The definitive version of MaPAct will be administered to a sample of 130 patients to evaluate the psychometric properties of MaPAct.

A complete Rasch analysis will be performed, along with an evaluation of internal consistency and test-retest reliability in a sub-sample of subjects.

Finally, since skeletal muscle weakness, reduced exercise capacity, slow gait and reduced physical activity levels are well-known systemic effects in COPD, in order to estimate MaPAct criterion validity with COPD status, the correlations between MaPAct with Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage (18), hospital admissions or exacerbations as defined by the GOLD and symptoms as derived by mMRC and CAT scales will be evaluated.

Time for completing the MaPAct will be also assessed. In order to provide an estimate of the reliability of the MaPAct to describe objective physical activity, in a sub group of 30 patients a metabolic holter (SenseWear armband - 48 hours) will be used to measure daily calories, number of steps and Metabolic Equivalents (METS) that will be correlated with the MapAct.

Timeline On day 1 of the study, all the COPD patients will perform medical evaluation (medical history, physical examination and history of COPD exacerbations within 12 month), pulmonary function tests, blood gas analysis and MaPAct. On the subsequent day, while 40 consecutive patients will complete again MaPAct (+ 24 h) for intrarater variability determination, all subjects will perform a 6-minute walking test (6MWT) and evaluate perceived exertion (CR-10; modified Borg Scale; 19). In all subjects modified Medical Research Council- (mMRC Dyspnea Index; 20, 21), and COPD Assessment Test (CAT, 22) will be carried on.

The GOLD spirometric classification will be used to determine the severity of the disease: mild COPD, forced expiratory volume in one second (FEV1) ≥80% predicted; moderate COPD, 50%≤FEV1<80% predicted; and severe-to-very severe COPD, FEV1<50% predicted.

Statistical analysis Internal consistency

The internal consistency of the MaPAct will be assessed by calculating:

1. Cronbach's coefficient alpha: the closer this is to 1.0 the greater the internal consistency of the items in the scale. An alpha of 0.8 is a reasonable goal. Rules of thumb are: "Alpha > 0.9 Excellent; > 0.8 Good; > 0.7 Acceptable" (23);
2. Item-remainder correlation through the Spearman's rank correlation (ρ) coefficient to examine the correlations between each item and the sum of the remaining items, omitting that item from the total: a Spearman coefficient ρ > 0.40 will be considered as the minimum value for satisfactory item-to-total correlation (24).

Reproducibility Reliability coefficient will be estimated with intraclass correlation coefficient (ICC). Expecting to obtain ICC values of about .90, with a 95% confidence interval (CI) of .20, at least 32 subjects are required (25).

Rasch Analysis For Rasch analysis, a sample size of more than 100 persons will estimate item difficulty with an alpha of 0.05 within ± 0.5 logits (26).

The steps of analysis will be as follows:

1. Rating scale diagnostic. We will investigate whether the rating scale is being used in the expected manner. We evaluated the response categories as suggested by Linacre (27).
2. Validity, assessed by evaluating the goodness of fit of the real data to the modelled data, to test if there were items that do not fit the model expectations. We will consider mean-square (MnSq) > 0.7 and < 1.3 as an indicator of acceptable fit (28). Items outside this range will be considered underacting (MnSq > 1.3, suggesting the presence of unexpectedly high variability), or overfitting (MnSq < 0.7, indicating a too predictable pattern).
3. Reliability, evaluated in terms of separation, defined as the ratio of the person (or item) "true" standard deviation to the error standard deviation (29). Item separation is used to verify the item hierarchy and reflects the number of "strata" of measures that are statistically discernible. A separation of 2.0 is considered good and sufficient to allow stratification into 3 groups (30). A related index is the reliability of these separation indexes, which provides the degree of confidence that can be placed in the reproducibility of these estimates; the value of the coefficient varies from 0 to 1 (values > 0.80 are considered good, and > 0.90 excellent) (31).
4. Principal component analysis (PCA) on the standardized residuals will be used to investigate:

4.1. The dimensionality of the scale. In this case "unidimensionality" assumes that, after the removal of the trait that the scale intended to measure (the "Rasch factor"), the residuals will be uncorrelated and normally distributed (i.e. there are no principal components). The following criteria will be used to determine whether additional factors are likely to be present in the residuals: at least 50% of the variance explained by the Rasch factor, eigenvalue of the first contrast smaller than 3, and variance explained by each contrast smaller than 5%.

4.2. The local independence of items. High correlation (> 0.30) of residuals for 2 items indicates that they may not be locally independent or that there is a subsidiary dimension in the measurement that is not accounted for by the main Rasch dimension (32).

Criterion validity Spearman's rank correlation (ρ) coefficient will be used to examine the correlations between the MaPAct and the COPD status as indicated by GOLD stage, CAT and mMRC scores. The effect size for the correlation is expected medium to high (r ~ 0.4). In order to detect departure from the hypothesis (i.e. small effect size, r <= .2), the sample size required is 130 subjects (alpha = 0.05, beta = 0.8, one sided test).

Comparison with Objective Physical Activity

Spearman's rank correlation (ρ) coefficient will be used to examine the correlations between the MaPAct and the daily calories, number of steps and METS as measured with the metabolic holter:

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis in stable state, able to read and to write, that accept to sign informed consent

Exclusion Criteria:

* will be excluded all patients that were hospitalized in the 30 days before evaluation, patients with degenerative neuromuscular diseases, subjects with motor disabilities limiting deambulation, subjects with memory or comprehension problems, with dementia, parkinson disease, cognitive impairment, and subject that do not give their consent for the participation to the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2019-07-02 (Estimated)

PRIMARY OUTCOMES:
Questionnaire validity | six months
  Numeric score

SECONDARY OUTCOMES:
Questionnaire reliability | six months
  Numeric score

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Spanevello, professor, Study Director — Insubria University
Locations (1):
- ICS Maugeri, Tradate, Va, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Demeyer H, Burtin C, Van Remoortel H, Hornikx M, Langer D, Decramer M, Gosselink R, Janssens W, Troosters T. Standardizing the analysis of physical activity in patients with COPD following a pulmonary rehabilitation program. Chest. 2014 Aug;146(2):318-327. doi: 10.1378/chest.13-1968. PMID 24603844
- [Background] Cindy Ng LW, Mackney J, Jenkins S, Hill K. Does exercise training change physical activity in people with COPD? A systematic review and meta-analysis. Chron Respir Dis. 2012 Feb;9(1):17-26. doi: 10.1177/1479972311430335. Epub 2011 Dec 22. PMID 22194629
- [Background] Pitta F, Troosters T, Probst VS, Spruit MA, Decramer M, Gosselink R. Quantifying physical activity in daily life with questionnaires and motion sensors in COPD. Eur Respir J. 2006 May;27(5):1040-55. doi: 10.1183/09031936.06.00064105. PMID 16707399
- [Background] Dobbels F, de Jong C, Drost E, Elberse J, Feridou C, Jacobs L, Rabinovich R, Frei A, Puhan MA, de Boer WI, van der Molen T, Williams K, Pinnock H, Troosters T, Karlsson N, Kulich K, Rudell K; PROactive consortium; PROactive consortium. The PROactive innovative conceptual framework on physical activity. Eur Respir J. 2014 Nov;44(5):1223-33. doi: 10.1183/09031936.00004814. Epub 2014 Jul 17. PMID 25034563